CLINICAL TRIAL: NCT01981005
Title: A PHASE 1, SINGLE-CENTER, OPEN-LABEL STUDY INVESTIGATING THE EXCRETION BALANCE, PHARMACOKINETICS AND METABOLISM OF A SINGLE ORAL DOSE AND PHARMACOKINETICS OF AN INTRAVENOUS TRACER OF [14-C]-RO5424802 IN HEALTHY MALE SUBJECTS
Brief Title: A Study of the Elimination, Pharmacokinetics, and Metabolism of RO5424802
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP28989
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — alectinib

ARMS (1):
- RO5424802 (Experimental)
  Interventions: Drug: RO5424802

INTERVENTIONS:
Drug: RO5424802 — Single oral doses followed by IV or oral administration of a 14C-labeled tracer

SUMMARY:
This non-randomized, single group, open-label study will investigate the mass balance, routes of elimination, pharmacokinetics, and metabolism of a single oral dose of RO5424802 and the pharmacokinetics of a 14C-labeled tracer in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male adults, 18 to 45 years of age, inclusive
* Body mass index (BMI) from 18 to 32 kg/m2, inclusive
* Willingness to use effective contraception as outlined in the protocol
* Willingness to abstain from alcohol and xanthine-containing beverages or food (coffee, tea, cola, chocolate and "energy drinks") from 72 hours prior to the first dose until discharged
* Willingness to avoid prolonged sun exposure and guard against sunburn during study & follow-up

Exclusion Criteria:

* Clinically significant medical history or findings in physical examination, vital signs, or laboratory test results prior to study start
* Positive screening tests for hepatitis B or C, HIV, alcohol, drugs of abuse, or tobacco
* Regular smoking within 6 months prior to first dosing. Subjects should avoid smoky environments for at least 1 week prior to each cotinine screen
* Excessive alcohol consumption
* Use of any metabolic inducers (including herbals such as St. John's Wort) within 4 weeks or 5 half-lives (whichever is longer) before the first dose of study medication, including but not limited to: rifampin, rifabutin, glucocorticoids, carbamazepine, phenytoin and phenobarbital
* Regular work with ionizing radiation or radioactive material
* Subjects enrolled in a previous radiolabel study or who have received radiotherapy within 12 months prior to first dosing such that total radioactivity over a 12 month period would exceed an acceptable radiation burden > 0.1 mSv
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work or participation in a medical trial in the previous year
* Strenuous activity, sunbathing, or contact sports are not allowed from 4 days prior to entry into the clinical site until study follow-up
* Participation in an investigational drug or device study within 60 days (or 6 months for biologic therapies) prior to first dosing

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Elimination: Amount of drug excreted in urine/feces over the study period | Days 11 to 15
Pharmacokinetics: Bioavailability (Area under the plasma concentration-time curve [AUC]) after administration of RO5424802 | Days 1 to 25

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | Days 1 to 25
Pharmacokinetics: Metabolite identification in plasma, urine, and feces. | Days 11 to 25

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands